CLINICAL TRIAL: NCT03691623
Title: A Randomised, Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics and Antiviral Activity of Multiple Doses of Orally Administered EDP-938 Against Respiratory Syncytial Virus Infection in the Virus Challenge Model.
Brief Title: A Phase 2a Study to Evaluate EDP-938 in the Virus Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: hVIVO Services Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 938-101
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2019-08

CONDITIONS: RSV Infection
Keywords: challenge study; RSV; antiviral; RSV-A Memphis 37b
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- EDP-938 Arm A (Experimental): Subjects will take EDP-938 Dose 1 oral suspension for 5 days
  Interventions: Drug: EDP-938 Dose 1
- EDP-938 Arm B (Experimental): Subjects will take EDP-938 Dose 2 oral suspension for 5 days
  Interventions: Drug: EDP-938 Dose 2
- Placebo Arm C (Placebo Comparator): Subjects will take matching placebo oral suspension for 5 days
  Interventions: Drug: Placebo
- EDP-938 Arm D (Experimental): Subjects will take EDP-938 Dose 3 oral suspension for 5 days
  Interventions: Drug: EDP-938 Dose 3
- EDP-938 Arm E (Experimental): Subjects will take EDP-938 Dose 4 oral suspension for 5 days
  Interventions: Drug: EDP-938 Dose 4
- Placebo Arm F (Placebo Comparator): Subjects will take matching placebo oral suspension for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-938 Dose 1 — Oral suspension for 5 days
  Arms: EDP-938 Arm A
Drug: EDP-938 Dose 2 — Oral suspension for 5 days
  Arms: EDP-938 Arm B
Drug: Placebo — Oral suspension for 5 days
  Arms: Placebo Arm C
Drug: EDP-938 Dose 3 — Oral suspension for 5 days
  Arms: EDP-938 Arm D
Drug: EDP-938 Dose 4 — Oral suspension for 5 days
  Arms: EDP-938 Arm E
Drug: Placebo — Oral suspension for 5 days
  Arms: Placebo Arm F

SUMMARY:
A randomised, Phase 2a, double-blind, placebo-controlled study to evaluate the safety, pharmacokinetics and antiviral activity of multiple doses of orally administered EDP-938 in healthy subjects infected with RSV-A Memphis 37b. This study is designed to compare the antiviral effect of EDP-938 compared to a placebo control in the respiratory syncytial virus challenge model.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject
* Age 18 to 55 years, inclusive
* In good health with no history of major medical conditions
* A total body weight ≥ 50 kg and Body Mass Index (BMI) ≥ 18 kg/m^2 and ≤ 30kg/m^2

Exclusion Criteria:

* Pregnant or nursing females
* Acute or chronic medical illness
* Abnormal lung function
* Positive for human immunodeficiency virus (HIV), active hepatitis A, B or C test
* Nose or nasopharynx abnormalities
* Receipt of any investigational drug within 3 months prior to the planned date of viral challenge/first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- hVIVO Services Limited (hVIVO), London, United Kingdom

REFERENCES:
- [Derived] Levene RE, DeVincenzo J, Conery AL, Ahmad A, Or YS, Rhodin MHJ. EDP-938 Has a High Barrier to Resistance in Healthy Adults Experimentally Infected with Respiratory Syncytial Virus. J Infect Dis. 2025 Feb 20;231(2):e290-e298. doi: 10.1093/infdis/jiae471. PMID 39441691
- [Derived] Ahmad A, Eze K, Noulin N, Horvathova V, Murray B, Baillet M, Grey L, Mori J, Adda N. EDP-938, a Respiratory Syncytial Virus Inhibitor, in a Human Virus Challenge. N Engl J Med. 2022 Feb 17;386(7):655-666. doi: 10.1056/NEJMoa2108903. PMID 35172056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 179 participants enrolled in the trial at one site in the United Kingdom from October 2018 to October 2019.
Pre-assignment Details: For Part 1, 115 participants were inoculated with respiratory syncytial virus-A (RSV-A) Memphis 37b and randomized, of whom 114 were treated. For Part 2, 64 participants were inoculated with RSV-A Memphis 37b of whom 63 were randomized and treated. The 178 randomized participants are included in the participant flow. One inoculated participant was not randomized to a specific treatment assignment and is not included in participant flow.
Groups:
- Part 1: EDP-938 600 mg: Participants were administered EDP-938 oral suspension of 600 mg followed after 12 hours by a placebo once daily (OD) for a total of 10 doses over 5 days.
- Part 1: EDP-938 500 mg Then 300 mg: Participants were administered EDP-938 oral suspension as a single loading dose of 500 mg followed after 12 hours by EDP-938 300 mg twice daily (BID) (every 12 hours) for a total of 10 doses over 5 days.
- Part 1: Placebo: Participants were administered a placebo BID (every 12 hours) for a total of 10 doses over 5 days.
- Part 2: EDP-938 600 mg Then 300 mg: Participants were administered a single loading dose of 600 mg EDP-938, followed by EDP-938 300 mg OD, and with dosing for 5 days.
- Part 2: EDP-938 400 mg Then 200 mg: Participants were administered a single loading dose of 400 mg EDP-938 followed by EDP-938 200 mg at 12 hours, then EDP-938 200 mg BID, and with dosing for 5 days.
- Part 2: Placebo: Participants were administered a placebo BID for 5 days, with dosing at 12 hour intervals.
Period: Overall Study
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Started | 39 | 38 | 38 | 21 | 21 | 21
Inoculated With Challenge Virus | 39 | 38 | 38 | 21 | 21 | 21
Received Treatment | 38 | 38 | 38 | 21 | 21 | 21
Completed | 39 | 38 | 38 | 21 | 21 | 21
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In Part 1, one participant in the Safety Analysis Set did not receive study treatment and is not included in this baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo | Total
Number analyzed (Participants) | 38 | 38 | 38 | 21 | 21 | 21 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 38 | 21 | 21 | 21 | 177
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 13 | 10 | 11 | 9 | 74
  Male | 25 | 20 | 25 | 11 | 10 | 12 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 1 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 1 | 0 | 4
  White | 33 | 32 | 31 | 18 | 17 | 19 | 150
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 3 | 2 | 2 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Respiratory Syncytial Virus (RSV) Viral Load
Description: Measured in nasal washes by quantitative reverse transcription polymerase chain reaction (RT-qPCR) in participants inoculated with respiratory syncytial virus-A (RSV-A) Memphis 37b.
Time Frame: Twice daily on Day 2 through Day 11 and once on Day 12
Population: Intent to Treat Infected (ITT-I) Analysis Set, defined as all randomised participants who received challenge virus and at least one dose of investigational medicinal product (IMP), and who met the criterion for laboratory confirmed respiratory syncytial virus (RSV) infection as per the definition of laboratory confirmed infection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*log10 copies/milliliter (mL)
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
hours*log10 copies/milliliter (mL) | 134.70 (85.1) | 113.51 (99.9) | 624.30 (51.7) | 80.61 (112.1) | 160.81 (63.3) | 808.28 (37.1)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -588.08, 95% CI 2-sided [-719.8 to -456.35]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -564.63, 95% CI 2-sided [-689.23 to -440.02]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -716.08, 95% CI 2-sided [-879.92 to -552.24]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -736.23, 95% CI 2-sided [-916.36 to -556.11]

2. Secondary Outcome: Area Under the Curve (AUC) of Total Symptom Score
Description: Total symptom scores (from the 10-item Diary Card) were used to calculate the AUC. Each individual symptom score was graded on a scale of 0-3, where Grade 0 is absence, Grade 1 is just noticeable, Grade 2 is bothersome but does not prevent participation in activities and Grade 3 is bothersome and interferes with activities:
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise (Tiredness)
  * Cough
  * Shortness of breath
  * Headache
  * Muscle/ joint ache/ stiffness
  Total symptom score is the sum of individual symptom scores with a potential range of 0 (best) to 30 (worst). Data presented is hours x score.
Time Frame: Three times daily on Day 0 to Day 11, once on Day 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*score
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
hours*score | 61.18 (347.8) | 37.36 (1640.1) | 252.49 (243.9) | 26.70 (730.2) | 27.81 (436.8) | 232.53 (530.9)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -355.91, 95% CI 2-sided [-506.12 to -205.69]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -326.64, 95% CI 2-sided [-469.68 to -183.6]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p = 0.001, ANCOVA; LS Mean Difference = -313.98, 95% CI 2-sided [-494.27 to -133.69]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p = 0.003, ANCOVA; LS Mean Difference = -312.73, 95% CI 2-sided [-508.05 to -117.4]

3. Secondary Outcome: Peak Total Symptom Score
Description: Peak total symptom score was defined as the highest total symptom score between first dose of study drug and Day 12. Values presented are a sum of individual symptom scores, with a potential range of 0 (best) to 30 (worst). Total symptom scores at the time of the first dose of study drug can be before or after dosing.
  Measured by the 10-item Diary Card. Each individual symptom score was graded on a scale of 0-3, where Grade 0 is absence, Grade 1 is just noticeable, Grade 2 is bothersome but does not prevent participation in activities and Grade 3 is bothersome and interferes with activities:
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise (Tiredness)
  * Cough
  * Shortness of breath
  * Headache
  * Muscle/ joint ache/ stiffness
Time Frame: Day 2 to Day 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Scores on a scale
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
Scores on a scale | 2.3 (53.9) | 1.9 (89.8) | 4.9 (77.9) | 1.6 (68.5) | 1.8 (55.6) | 4.2 (85.8)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.7, 95% CI 2-sided [-5.3 to -2]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.9, 95% CI 2-sided [-5.5 to -2.4]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = -3, 95% CI 2-sided [-4.9 to -1.2]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p = 0.006, ANCOVA; LS Mean Difference = -2.9, 95% CI 2-sided [-4.9 to -0.9]

4. Secondary Outcome: Total Symptom Score
Description: Measured by the 10-item Diary Card. Each individual symptom score was graded on a scale of 0-3, where Grade 0 is absence, Grade 1 is just noticeable, Grade 2 is bothersome but does not prevent participation in activities and Grade 3 is bothersome and interferes with activities. Total symptom score is the sum of individual symptom scores with a potential range of 0 (best) to 30 (worst).
  * Runny nose
  * Stuffy nose
  * Sneezing
  * Sore throat
  * Earache
  * Malaise (Tiredness)
  * Cough
  * Shortness of breath
  * Headache
  * Muscle/ joint ache/ stiffness
Time Frame: Day 2 to Day 9
Population: Intent to Treat Infected (ITT-I) Analysis Set, defined as all randomised participants who received challenge virus and at least one dose of investigational medicinal product (IMP), and who met the criterion for laboratory confirmed respiratory syncytial virus (RSV) infection as per the definition of laboratory confirmed infection. For cases of 0 participants analyzed, data were not collected from any participants for that time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Scores on a scale
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
Scores on a scale
  Relative Day 2 Assessment 1: number analyzed (Participants) | 25 | 31 | 29 | 15 | 11 | 12
  Relative Day 2 Assessment 1 | 0.9 (97.5) | 0.8 (155.4) | 1.9 (117.0) | 0.5 (140.8) | 0.3 (222.5) | 3.0 (66.6)
  Relative Day 2 Assessment 2 | 0.8 (94.0) | 0.7 (160.3) | 2.4 (110.3) | 0.4 (185.2) | 0.5 (179.8) | 2.9 (82.5)
  Relative Day 2 Assessment 3 | 0.5 (117.0) | 0.6 (184.4) | 2.7 (94.9) | 0.3 (196.2) | 0.2 (331.7) | 2.6 (94.3)
  Relative Day 3 Assessment 1 | 0.4 (137.3) | 0.7 (148.5) | 2.6 (99.1) | 0.4 (166.9) | 0.2 (254.2) | 2.2 (103.0)
  Relative Day 3 Assessment 2 | 0.4 (144.3) | 0.6 (175.2) | 2.7 (90.5) | 0.3 (207.0) | 0.3 (237.1) | 2.3 (101.0)
  Relative Day 3 Assessment 3 | 0.3 (190.9) | 0.6 (167.7) | 2.5 (103.7) | 0.2 (332.6) | 0.3 (276.4) | 2.2 (95.3)
  Relative Day 4 Assessment 1 | 0.3 (177.1) | 0.5 (154.9) | 2.3 (103.8) | 0.2 (343.9) | 0.2 (254.2) | 1.9 (92.6)
  Relative Day 4 Assessment 2 | 0.3 (186.5) | 0.6 (163.1) | 1.8 (115.3) | 0.1 (387.3) | 0.1 (331.7) | 1.7 (85.0)
  Relative Day 4 Assessment 3 | 0.3 (263.0) | 0.4 (163.5) | 1.8 (103.1) | 0.2 (280.3) | 0.1 (331.7) | 1.8 (88.3)
  Relative Day 5 Assessment 1 | 0.2 (228.2) | 0.5 (158.9) | 1.6 (108.3) | 0.2 (244.9) | 0.2 (254.2) | 1.6 (87.9)
  Relative Day 5 Assessment 2 | 0.3 (191.3) | 0.4 (177.1) | 1.4 (109.2) | 0.2 (314.0) | 0.2 (254.2) | 1.4 (112.8)
  Relative Day 5 Assessment 3 | 0.1 (364.8) | 0.4 (162.0) | 1.3 (115.9) | 0.1 (280.3) | 0.1 (331.7) | 1.4 (89.6)
  Relative Day 6 Assessment 1 | 0.2 (300.9) | 0.4 (186.9) | 1.2 (106.0) | 0.2 (314.0) | 0.2 (237.1) | 1.5 (83.3)
  Relative Day 6 Assessment 2 | 0.2 (288.7) | 0.4 (186.9) | 1.0 (112.8) | 0.1 (387.3) | 0.3 (185.4) | 1.2 (102.4)
  Relative Day 6 Assessment 3: number analyzed (Participants) | 22 | 23 | 24 | 15 | 10 | 11
  Relative Day 6 Assessment 3 | 0.2 (280.9) | 0.3 (184.6) | 1.0 (100.5) | 0.1 (387.3) | 0.1 (210.8) | 1.1 (116.5)
  Relative Day 7 Assessment 1: number analyzed (Participants) | 22 | 23 | 24 | 15 | 10 | 11
  Relative Day 7 Assessment 1 | 0.2 (225.1) | 0.2 (205.3) | 0.7 (124.9) | 0.1 (387.3) | 0.1 (316.2) | 0.8 (126.1)
  Relative Day 7 Assessment 2: number analyzed (Participants) | 21 | 21 | 23 | 12 | 9 | 11
  Relative Day 7 Assessment 2 | 0.2 (196.2) | 0.2 (162.0) | 0.7 (115.7) | 0.1 (346.4) | 0.1 (300.0) | 0.9 (153.5)
  Relative Day 7 Assessment 3: number analyzed (Participants) | 18 | 17 | 19 | 11 | 7 | 10
  Relative Day 7 Assessment 3 | 0.2 (291.0) | 0.2 (185.8) | 0.9 (89.9) | 0.1 (331.7) | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.7 (179.2)
  Relative Day 8 Assessment 1: number analyzed (Participants) | 18 | 17 | 19 | 11 | 7 | 10
  Relative Day 8 Assessment 1 | 0.1 (291.0) | 0.2 (199.9) | 0.9 (94.9) | 0.1 (331.7) | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.5 (153.7)
  Relative Day 8 Assessment 2: number analyzed (Participants) | 14 | 13 | 17 | 7 | 4 | 7
  Relative Day 8 Assessment 2 | 0.1 (374.2) | 0.1 (244.1) | 0.9 (99.4) | 0.2 (264.6) | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.2 (170.8)
  Relative Day 8 Assessment 3: number analyzed (Participants) | 5 | 5 | 10 | 4 | 0 | 4
  Relative Day 8 Assessment 3 | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.4 (149.1) | 0.6 (129.1) | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 |  | 0.2 (200.0)
  Relative Day 9 Assessment 1: number analyzed (Participants) | 5 | 5 | 10 | 4 | 0 | 4
  Relative Day 9 Assessment 1 | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.4 (140.5) | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 |  | 0.2 (200.0)
  Relative Day 9 Assessment 2: number analyzed (Participants) | 3 | 3 | 5 | 4 | 0 | 2
  Relative Day 9 Assessment 2 | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 | 0.5 (91.3) | 0.0 (NA) — %CV not calculable as Geometric Mean = 0.0 |  | 0.4 (141.4)

5. Secondary Outcome: Time to Peak Total Symptom Score
Description: Time to peak total symptom score was defined as the time in days to the highest total symptom score between first dose of study drug and Day 12. Total symptom scores at the time of the first dose of study drug can be before or after dosing.
Time Frame: Day 2 to Day 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
Days | 1.18 (137.8) | 1.76 (110.0) | 2.15 (71.4) | 1.45 (131.9) | 1.09 (136.4) | 1.94 (80.5)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p = 0.199, ANCOVA; LS Mean Difference = -0.82, 95% CI 2-sided [-2.09 to 0.44]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p = 0.714, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.98 to 1.43]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p = 0.844, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-2.15 to 1.77]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p = 0.21, ANCOVA; LS Mean Difference = -1.34, 95% CI 2-sided [-3.46 to 0.79]

6. Secondary Outcome: Time to Resolution From Peak Total Symptom Score
Description: Time to resolution from peak total symptom score was defined as the time in days from the highest total symptom score (between first dose of study drug and Day 12) until the start of the first 24-hour symptom-free period (after the highest total symptom score). Total symptom scores at the time of the first dose of study drug can be before or after dosing.
Time Frame: Day 2 to Day 12
Population: Intent to Treat Infected (ITT-I) Analysis Set, defined as all randomised participants who received challenge virus and at least one dose of investigational medicinal product (IMP), and who met the criterion for laboratory confirmed respiratory syncytial virus (RSV) infection as per the definition of laboratory confirmed infection.
  9 participants in Part 1 and 5 participants in Part 2 were excluded from the analysis due to having no symptoms in the interval first dose of study drug to Day 12.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 23 | 24 | 30 | 12 | 10 | 11
Days | 2.49 (70.1) | 2.83 (77.5) | 3.30 (61.7) | 2.19 (70.0) | 1.38 (116.5) | 5.17 (383)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p = 0.145, ANCOVA; LS Mean Difference = -1.01, 95% CI 2-sided [-2.37 to 0.36]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p = 0.352, ANCOVA; LS Mean Difference = -0.65, 95% CI 2-sided [-2.03 to 0.73]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p = 0.002, ANCOVA; LS Mean Difference = -2.85, 95% CI 2-sided [-4.55 to -1.15]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.4, 95% CI 2-sided [-5.19 to -1.61]

7. Secondary Outcome: Total Weight of Nasal Mucus Produced
Description: Measured via weighed paper tissues and reported as a mean total across all study days.
Time Frame: Day 2 to Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
Grams | 12.965 (13.0314) | 7.428 (11.1324) | 33.416 (37.8072) | 2.983 (4.4226) | 4.716 (6.0015) | 22.391 (20.6005)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -24.081, 95% CI 2-sided [-36.554 to -11.607]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -25.954, 95% CI 2-sided [-37.695 to -14.213]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -18.13, 95% CI 2-sided [-27.176 to -9.083]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -19.329, 95% CI 2-sided [-29.106 to -9.552]

8. Secondary Outcome: Peak Viral Load
Description: Peak viral load was defined as the highest quantitative reverse transcription polymerase chain reaction (RT-qPCR) viral load value between first dose of study drug and Day 12. Measured by nasal wash RT-qPCR.
Time Frame: Day 2 to Day 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 copies/milliliter (mL)
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
log10 copies/milliliter (mL) | 4.3552 (1.56334) | 4.3111 (1.76974) | 6.4727 (1.60659) | 3.9718 (1.78873) | 4.7727 (1.35014) | 7.0973 (1.24388)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.1292, 95% CI 2-sided [-2.8491 to -1.4093]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.1129, 95% CI 2-sided [-2.7938 to -1.4319]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.2191, 95% CI 2-sided [-4.1915 to -2.2467]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.7831, 95% CI 2-sided [-3.8522 to -1.714]

9. Secondary Outcome: Time to Peak Viral Load
Description: Time to peak viral load was defined as the time to the highest quantitative reverse transcription polymerase chain reaction (RT-qPCR) viral load value between first dose of study drug and Day 12. Measured by nasal wash RT-qPCR.
Time Frame: Day 2 to Day 12
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 31 | 30 | 15 | 11 | 12
Days | 0.74 (75.6) | 0.80 (130.2) | 2.59 (48.5) | 0.88 (181.3) | 0.79 (64.0) | 3.43 (33.7)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.01, 95% CI 2-sided [-2.67 to -1.35]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.78, 95% CI 2-sided [-2.4 to -1.16]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p = 0.009, ANCOVA; LS Mean Difference = -1.98, 95% CI 2-sided [-3.43 to -0.54]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p = 0.004, ANCOVA; LS Mean Difference = -2.41, 95% CI 2-sided [-4 to -0.82]

10. Secondary Outcome: Time to Resolution From Peak Viral Load
Description: Time to resolution from peak viral load was defined as the time from peak until first confirmed undetectable assessment between first dose of study drug and Day 12. Measured by by nasal wash quantitative reverse transcription polymerase chain reaction (RT-qPCR).
Time Frame: Day 2 to Day 12
Population: Intent to Treat Infected (ITT-I) Analysis Set, defined as all randomised participants who received challenge virus and at least one dose of investigational medicinal product (IMP), and who met the criterion for laboratory confirmed respiratory syncytial virus (RSV) infection as per the definition of laboratory confirmed infection. Participants were excluded from the analysis if it was concluded that the criteria for laboratory-confirmed RSV infection were not met.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 30 | 30 | 14 | 11 | 12
Days | 2.03 (72.1) | 2.02 (79.7) | 4.03 (47.5) | 1.67 (77.1) | 1.63 (43.7) | 3.58 (45.6)
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.1, 95% CI 2-sided [-3.04 to -1.17]
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2, 95% CI 2-sided [-2.89 to -1.11]
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -1.97, 95% CI 2-sided [-3.06 to -0.89]
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -2.46, 95% CI 2-sided [-3.64 to -1.29]

11. Secondary Outcome: Time to Cessation of Virus Detection
Description: Time to cessation of virus detection was measured by nasal wash quantitative reverse transcription polymerase chain reaction (RT-qPCR).
Time Frame: Day 2 to Day 12
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 25 | 30 | 30 | 14 | 11 | 12
Days | 3.5 [2.0 to 4.5] | 3.2 [1.5 to 4.5] | 8.5 [6.5 to NA] — Upper quartile is non-estimable as there were too many censored values in the placebo group. If a participant did not have a confirmed undetectable assessment after their peak, the time to cessation was censored (at the last detectable RT-qPCR result). | 2.7 [1.5 to 4.0] | 2.5 [1.5 to 3.5] | 8.5 [7.0 to 9.0]
Statistical Analysis 1: Comparison: Part 1: EDP-938 600 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 2: Comparison: Part 1: EDP-938 500 mg Then 300 mg vs Part 1: Placebo; Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 3: Comparison: Part 2: EDP-938 600 mg Then 300 mg vs Part 2: Placebo; Test type: Superiority; p = 0.001, Log Rank
Statistical Analysis 4: Comparison: Part 2: EDP-938 400 mg Then 200 mg vs Part 2: Placebo; Test type: Superiority; p < 0.001, Log Rank

12. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any untoward medical occurrence in participants that happened after study drug administration. Any clinically significant physical examinations, vital signs, clinical laboratory tests (including biochemistry, hematology, coagulation [if required], cardiac enzymes and urine analysis), 12-lead electrocardiograms (ECGs) and spirometry results were recorded as adverse events.
Time Frame: Day 2 to Day 28
Population: Safety Analysis Set, defined as all participants who received challenge virus, whether they received study drug or not. One inoculated participant was not randomized to a specific treatment assignment and is not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
Number analyzed (Participants) | 38 | 38 | 38 | 21 | 21 | 21
Participants | 20 | 21 | 21 | 8 | 10 | 11

13. Secondary Outcome: Maximum Plasma Concentration (Cmax) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: Day 2: pre-dose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10 and 12 hours post-dose; and Day 7: 15, 24, 30, 36, 48, 60, and 72 hours post-dose
Population: Pharmacokinetic (PK) Analysis Set, defined as all Intent to Treat (ITT) participants with at least one post-dose PK result. Participants were excluded from the analysis if plasma concentrations were below the limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 37 | 21 | 20
nanograms per milliliter (ng/mL)
  EDP-938 First Dose | 1370 (49.7) | 1151 (46.9) | 1237.91 (33.2) | 800.73 (44.9)
  EDP-938 Last Dose | 1740 (52.8) | 1480 (33.4) | 1010 (15.9) | 901 (27.9)
  EP-024636 First Dose | 256 (39.3) | 215 (41.3) | 264 (42.0) | 177 (48.2)
  EP-024636 Last Dose | 361 (34.8) | 342 (27.8) | 230 (23.0) | 232 (32.0)
  EP-024594 First Dose | 96.3 (48.1) | 76.8 (54.8) | 102 (61.1) | 72.3 (49.1)
  EP-024594 Last Dose | 203 (32.6) | 240 (30.1) | 130 (44.1) | 168 (32.9)
  EP-024595 First Dose | 150 (63.2) | 102 (79.6) | 167 (81.1) | 100 (72.1)
  EP-024595 Last Dose | 717 (45.6) | 1000 (49.1) | 499 (89.0) | 692 (50.5)

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 37 | 21 | 20
Hours
  EDP-938 First Dose | 4.56 [2.0 to 10.0] | 5.00 [1.0 to 12.0] | 5.80 [1.9 to 10.2] | 6.07 [2.0 to 10.2]
  EDP-938 Last Dose | 4.52 [1.9 to 17.0] | 4.10 [0.0 to 10.1] | 4.98 [1.0 to 15.9] | 4.04 [0.0 to 10.0]
  EP-024636 First Dose | 5.91 [2.9 to 23.5] | 5.97 [2.0 to 12.0] | 7.97 [3.1 to 11.9] | 6.99 [2.0 to 11.8]
  EP-024636 Last Dose | 5.00 [2.8 to 15.0] | 4.88 [0.5 to 8.0] | 6.00 [3.0 to 17.0] | 4.04 [0.0 to 8.3]
  EP-024594 First Dose | 10.07 [4.1 to 24.1] | 10.23 [4.0 to 12.0] | 11.83 [6.2 to 23.8] | 10.14 [4.9 to 11.9]
  EP-024594 Last Dose | 8.07 [4.0 to 20.1] | 4.98 [0.0 to 12.0] | 8.00 [0.5 to 17.2] | 5.03 [0.0 to 8.3]
  EP-024595 First Dose | 23.72 [8.0 to 24.1] | 11.85 [8.0 to 12.2] | 23.75 [11.8 to 24.0] | 11.83 [5.8 to 12.0]
  EP-024595 Last Dose | 10.90 [3.0 to 22.0] | 5.07 [0.4 to 12.0] | 11.88 [2.8 to 22.3] | 4.04 [0.0 to 9.9]

15. Secondary Outcome: Terminal Phase Half-Life (t1/2) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: Day 2 and Day 6: Pre-dose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post-dose; Day 7 only: 15, 24, 30, 36, 48, 60, and 72 hours post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 35 | 21 | 20
Hours
  EDP-938 | 14.5 (25.4) | 13.8 (27.4) | 14.5 (31.3) | 13.7 (23.5)
  EP-024636 | 14.5 (21.5) | 13.4 (21.1) | 14.4 (29.8) | 13.5 (21.2)
  EP-024594 | 17.8 (18.2) | 16.2 (18.5) | 17.5 (25.1) | 15.4 (17.0)
  EP-024595 | 28.5 (38.2) | 25.5 (25.1) | 22.7 (15.6) | 23.0 (19.4)

16. Secondary Outcome: Apparent Systemic Clearance at Steady State (CLss/F) of EDP-938
Time Frame: as for outcome 15
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litres per hour
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 35 | 21 | 20
litres per hour | 26.9 (44.8) | 24.1 (28.4) | 21.3 (17.6) | 25.0 (23.9)

17. Secondary Outcome: Terminal Phase Rate Constant Calculated by Linear Regression of the Terminal Loglinear Portion of the Concentration vs. Time Curve (λz) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: as for outcome 15
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 35 | 21 | 20
1/hour
  EDP-938 | 0.05 (1.2) | 0.05 (1.6) | 0.05 (1.5) | 0.05 (1.2)
  EP-024636 | 0.05 (1.1) | 0.05 (1.2) | 0.05 (1.3) | 0.05 (1.1)
  EP-024594 | 0.04 (0.7) | 0.04 (0.8) | 0.04 (1.0) | 0.05 (0.8)
  EP-024595 | 0.03 (1.3) | 0.03 (0.9) | 0.03 (0.5) | 0.03 (0.6)

18. Secondary Outcome: Volume of Distribution at Steady State (Vss/F) of EDP-938
Time Frame: as for outcome 15
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre(s)
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 35 | 21 | 20
litre(s) | 560 (42.8) | 476 (23.1) | 442 (24.1) | 491 (28.8)

19. Secondary Outcome: Plasma Concentration at 12 Hours (C12) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: Day 2 and Day 7; 12 hours post-dose
Population: Pharmacokinetic (PK) Analysis Set, defined as all Intent to Treat (ITT) participants with at least one post-dose PK result. Participants were excluded from the analysis if plasma concentrations were below the limit of quantification. C12 is only reported for twice daily (BID) dosing groups relative to the last dose. Data were specifically collected for BID dosing groups at the specified times.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 0 | 37 | 0 | 20
nanograms per milliliter (ng/mL)
  EDP-938 First Dose |  | 679.35 (34.5) |  | 565.60 (39.5)
  EDP-938 Last Dose |  | 822 (35.2) |  | 525 (30.0)
  EP-024636 First Dose |  | 168 (32.1) |  | 149 (41.0)
  EP-024636 Last Dose |  | 228 (27.8) |  | 153 (28.9)
  EP-024594 First Dose |  | 75.3 (54.4) |  | 68.8 (50.8)
  EP-024594 Last Dose |  | 188 (27.4) |  | 133 (31.7)
  EP-024595 First Dose |  | 100 (79.6) |  | 99.3 (75.4)
  EP-024595 Last Dose |  | 705 (39.1) |  | 515 (40.2)

20. Secondary Outcome: Plasma Concentration at 24 Hours (C24) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: Day 2 and Day 7; 24 hours post-dose
Population: Pharmacokinetic (PK) Analysis Set, defined as all Intent to Treat (ITT) participants with at least one post-dose PK result. Participants were excluded from the analysis if plasma concentrations were below the limit of quantification. C24 is only reported for once daily (OD) dosing groups relative to last dose. Data were specifically collected for OD dosing groups at the specified times.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 37 | 0 | 21 | 0
nanograms per milliliter (ng/mL)
  EDP-938 First Dose | 404 (46.9) |  | 453 (31.6) |
  EDP-938 Last Dose | 491 (56.4) |  | 287 (74.0) |
  EP-024636 First Dose | 121 (43.5) |  | 136 (30.5) |
  EP-024636 Last Dose | 148 (44.4) |  | 88.3 (64.8) |
  EP-024594 First Dose | 78.8 (43.7) |  | 87.8 (56.0) |
  EP-024594 Last Dose | 127 (29.3) |  | 74.5 (72.4) |
  EP-024595 First Dose | 142 (57.5) |  | 163 (79.4) |
  EP-024595 Last Dose | 461 (41.6) |  | 287 (93.8) |

21. Secondary Outcome: Area Under the Concentration Time Curve Time 0 to Time of Last Quantifiable Concentration (AUC0-last) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 37 | 21 | 20
ng*hr/mL
  EDP-938 First Dose | 16730 (47.0) | 7540 (45.8) | 16420 (24.0) | 5970 (40.5)
  EDP-938 Last Dose | 32000 (52.9) | 27300 (40.8) | 20500 (32.1) | 17800 (29.0)
  EP-024636 First Dose | 3800 (42.9) | 1490 (49.3) | 4080 (36.2) | 1300 (45.9)
  EP-024636 Last Dose | 8680 (42.9) | 7690 (32.8) | 5550 (24.1) | 5180 (28.8)
  EP-024594 First Dose | 1610 (55.3) | 512 (73.1) | 1740 (64.2) | 487 (51.5)
  EP-024594 Last Dose | 6880 (31.7) | 7160 (27.5) | 4320 (37.3) | 4990 (31.6)
  EP-024595 First Dose | 2510 (72.1) | 540 (95.6) | 2420 (83.1) | 541 (67.1)
  EP-024595 Last Dose | 29600 (40.5) | 36900 (38.4) | 19700 (77.1) | 25800 (46.6)

22. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Over the Dosing Interval (AUC0-tau) of EDP-938 and Its Metabolites
Description: The metabolites of EDP-938 that were assessed were EP-024636, EP-024594 and EP-024595.
Time Frame: as for outcome 15
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 35 | 21 | 20
ng*hr/mL
  EDP-938 | 22300 (46.5) | 12500 (29.7) | 14100 (18.5) | 8010 (24.9)
  EP-024636 | 5770 (36.1) | 3270 (25.2) | 3640 (24.5) | 2210 (30.8)
  EP-024594 | 3830 (30.6) | 2470 (26.1) | 2410 (45.4) | 1710 (33.8)
  EP-024595 | 12100 (41.9) | 8950 (36.7) | 8350 (82.0) | 6210 (44.3)

23. Secondary Outcome: Number of Participants With Correlation of Plasma Pharmacokinetic (PK) Area Under the Curve (AUC) and Viral Load AUC
Description: The overall criteria to define correlation was based on identifying a PK AUC associated with a less favorable viral load AUC i.e. a low PK AUC and a high viral load AUC indicated a correlation.
Time Frame: Day 2 to Day 18
Population: Pharmacokinetic (PK) Analysis Set, defined as all Intent to Treat (ITT) participants with at least one post-dose PK result.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 38 | 21 | 21
Participants | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants With Correlation of Plasma Pharmacokinetic (PK) Area Under the Curve (AUC) and Total Symptom Score (TSS) AUC
Description: The overall criteria to define correlation was based on identifying a PK AUC associated with a less favorable TSS AUC, i.e. a low PK AUC and a high TSS AUC indicated a correlation.
Time Frame: Day 2 to Day 18
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg
Number analyzed (Participants) | 38 | 38 | 21 | 21
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality was monitored from enrollment until end of study (Day 28) for the safety analysis population which included all participants who received challenge virus, regardless of whether they received study drug or not. Treatment-emergent serious and other adverse events (AEs) were monitored from Day 2 to Day 28 and only included participants in the safety analysis population who received study drug.
Description: An adverse event (AE) was defined as any untoward medical occurrence in participants (any unfavourable and unintended sign [including an abnormal laboratory finding], symptom, or disease temporally associated with the investigational medicinal product [IMP], whether or not considered related to IMP, or for Human Viral Challenge studies, the Challenge Virus). AEs were recorded in the source documents as they are reported, whether volunteered by a participant or in response to questioning.
Arm/Group | Part 1: EDP-938 600 mg | Part 1: EDP-938 500 mg Then 300 mg | Part 1: Placebo | Part 2: EDP-938 600 mg Then 300 mg | Part 2: EDP-938 400 mg Then 200 mg | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38 | 0/38 | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 20/38 | 21/38 | 21/38 | 8/21 | 10/21 | 11/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: EDP-938 600 mg (N=38) | Part 1: EDP-938 500 mg Then 300 mg (N=38) | Part 1: Placebo (N=38) | Part 2: EDP-938 600 mg Then 300 mg (N=21) | Part 2: EDP-938 400 mg Then 200 mg (N=21) | Part 2: Placebo (N=21)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEV1/FVC ratio decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forced vital capacity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of Sponsor Data shall be made by Sponsor with input from principal investigator (PIs). If no publication within 24 months after study completion, PI may publish Sponsor Data with sponsor's prior written consent. Prior to submitting or presenting data, Sponsor has at least 60 days to to review and comment.

DOCUMENTS (2):
  • Study Protocol (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03691623/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03691623/SAP_001.pdf